CLINICAL TRIAL: NCT02900573
Title: Caregivers Confronted With the Withdrawal of Artificial Nutrition at the End of Life: Perception and Experienced Difficulties
Brief Title: Withdrawal of Artificial Nutrition at the End of Life (PERCEPAL)
Acronym: PERCEPAL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-01Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-08

CONDITIONS: Palliative Care Nursing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Withdrawing artificial nutrition in palliative care is an issue that often leads to ethical dilemmas among health care providers, despite clinical guidelines.

DETAILED DESCRIPTION:
The benefit of artificial nutrition in terminally ill patients has been a highly debated issue for the past 30 years, and abundant data are available regarding its effects on patients. Several clinical guidelines have specified the criteria to be considered before initiating artificial nutrition or hydration. If these guidelines appear consensual in theory, the situation is much less straightforward in practice. The attitude of physicians appeared very variable when it came to prescribing or withholding artificial nutrition or hydration, and the lack of training, among other parameters, seemingly encouraged health care professionals to prescribe artificial nutrition or hydration. Furthermore, the decision of the care provider is unconsciously complicated due to figurative representations associated with food regarding, among other aspects, the mother-child relationship, social cohesion, or religious beliefs.

These differences are more important since the opinion of physicians and nurses is the one that carries the most influence on the patients' decision when deciding to initiate artificial nutrition and because artificial nutrition and hydration are a common source of ethical dilemmas in health care teams. Furthermore, stopping artificial nutrition or hydration could be misconstrued as euthanasia.

ELIGIBILITY:
Inclusion Criteria:

* nurses, and nurses' aides working in medicine, surgery, and palliative care departments of the regional hospital of Metz-Thionville

Exclusion Criteria:

* Care providers working in pediatrics, gynecology and obstetrics, psychiatry, and emergency departments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Senior nurses (which are not directly in contact with the patient but involved in team management), nurses (which perform patient care), and nurses' aides (which are involved in hygiene measures) working in the medicine, surgery, and palliative care departments of the regional hospital of Metz-Thionville.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Experience of health care providers confronted with the withdrawing of artificial nutrition at the end of life | month 4
  Cross-sectional survey questionnaire

SECONDARY OUTCOMES:
Experienced difficulties | month 4
  Cross-sectional survey questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Benoît LEHEUP, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No